CLINICAL TRIAL: NCT04249934
Title: The Effects of Caffeine on DIEP Flap Perfusion: A Pilot Study
Brief Title: The Effects of Caffeine on Deep Inferior Epigastric Perforator (DIEP) Flap Perfusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to restrictions related to patient care secondary to covid pandemic.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Adeyiza Momoh, Associate Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUM00142366
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Breast Reconstruction; Deep Inferior Epigastric Perforator; Microvascular Free Flap Transfer

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient and observer will be blinded to which group they were assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeinated Coffee (Experimental)
  Interventions: Dietary Supplement: Caffeinated Coffee
- Decaffeinated Coffee (Active Comparator)
  Interventions: Dietary Supplement: DecaffeinatedCoffee

INTERVENTIONS:
Dietary Supplement: Caffeinated Coffee — A single 8 ounce cup of regular starbucks coffee will be given to the participant in the am post operative day two. Participants will have 15 minutes to consume the coffee. Additionally, medical record data will be collected up to 30 days after surgery.
  Arms: Caffeinated Coffee
Dietary Supplement: DecaffeinatedCoffee — A single 8 ounce cup of decaffeinated starbucks coffee will be given to the participant in the am post operative day two. Participants will have 15 minutes to consume the coffee. Additionally, medical record data will be collected up to 30 days after surgery.
  Arms: Decaffeinated Coffee

SUMMARY:
Women that require breast reconstruction and meet eligibility will be enrolled in this study. The study is being completed to determine the effect of caffeine in deep inferior epigastric perforator (DIEP) flap perfusion using the Vioptix tissue oximeter monitor and to determine if caffeine in the acute postoperative period affects overall flap complication or loss (complete loss from anastomotic issue).

The researchers hypothesize that a single 8 ounce cup of regular coffee will not affect free flap perfusion as indicated by the Vioptix, and that it will not affect overall free flap survival at thirty days.

ELIGIBILITY:
Inclusion Criteria:

* regular caffeine consumers undergoing unilateral or bilateral microsurgical breast reconstruction with DIEP flap(s) at the University of Michigan Health System

Exclusion Criteria:

* smokers
* hepatic or renal disease (comorbidities that affect caffeine metabolism)
* male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only women scheduled to undergo unilateral or bilateral microsurgical breast reconstruction will be enrolled
Enrollment: 0 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Analysis of feasibility | approximately 6 months after recruitment starts
  The total number of patients recruited per month, the rate of successful enrollment, and the rate of successful study completion will be evaluated.
Absolute value of tissue oxygenation saturation (StO2) | up to 165 minutes (30 minutes prior to coffee consumption, 15 minutes for coffee consumption, 120 more minutes after consumption)
  St02 will be measured using the Vioptix tissue oximeter monitor. These will be summarized using means and standard deviations.
Absolute value of tissue oxygenation saturation (StO2) rate of change | up to 165 minutes (30 minutes prior to coffee consumption, 15 minutes for coffee consumption, 120 more minutes after consumption)
  St02 will be measured using the Vioptix tissue oximeter monitor. These will be summarized using means and standard deviations.
Absolute value of tissue oxygenation saturation (StO2) amount of change | up to 165 minutes (30 minutes prior to coffee consumption, 15 minutes for coffee consumption, 120 more minutes after consumption)
  St02 will be measured using the Vioptix tissue oximeter monitor. These will be summarized using means and standard deviations.

SECONDARY OUTCOMES:
Incidence of minor flap complications in the caffeine and non-caffeine groups | up to 30 days post-operatively
  The complications will include delayed wound healing, wound dehiscence, hematoma, seroma formation, and infections requiring antibiotics.
Incidence of major flap complications in the caffeine and non-caffeine groups | up to 30 days post-operatively
  These complications will include any event that results in an unplanned trip to the operating room (e.g. arterial or venous thrombosis), and flap loss (e.g. flap failure, flap death).

CONTACTS AND LOCATIONS:
Overall Officials: Adeyiza Momoh, MD, Principal Investigator — University of Michigan; Theodore A Kung, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No